CLINICAL TRIAL: NCT05666804
Title: A 60-week, Phase IIIb, Randomized, Multi-center Study Assessing the Efficacy and Safety of a Personalized Monotherapy Regimen of Brolucizumab in Patients With Symptomatic Macular Polypoidal Choroidal Vasculopathy (PROUD Study)
Brief Title: Study Assessing the Efficacy and Safety of a Personalized Monotherapy Regimen of Brolucizumab in Patients With Symptomatic Macular Polypoidal Choroidal Vasculopathy
Acronym: PROUD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRTH258AKR03
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Macular Polypoidal Choroidal Vasculopathy (PCV)
Keywords: Neovascular age-related macular degeneration; polypoidal choroidal vasculopathy; anti-vascular endothelial growth factor; brolucizumab; personalized regimen; treat-and-extend; Retina damage; Retinal disease; Vascular disease; Eye disease; blind spot; fluid leak into or under the retina; blood leak into or under the retina; macular polypoidal choroidal vasculopathy (PCV); PCV
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy; Retinal Diseases; Vascular Diseases; Eye Diseases; Scotoma | interventions — brolucizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized regimen arm (Experimental): 1~3 x 4-week loading injections and one 8-week injection, followed by Treat-and-extend (T&E) regimen up to Week 56
  Interventions: Drug: Brolucizumab 6mg
- Standard regimen arm (Active Comparator): 3 x 4-week loading injections and disease activity assessment at week 16 followed by q12w/q8w up to Week 56
  Interventions: Drug: Brolucizumab 6mg

INTERVENTIONS:
Drug: Brolucizumab 6mg — Brolucizumab 6mg (intravitreal) Personalized regimen arm: 1~3 x 4-week loading injections and one 8-week injection, followed by Treat-and-extend (T&E) regimen up to Week 56
  Other Names: Beovu
  Arms: Personalized regimen arm
Drug: Brolucizumab 6mg — Brolucizumab 6mg(intravitreal) Standard q12w/q8w regimen arm: 3 x 4-week loading injections and disease activity assessment at week 16 followed by q12w/q8w up to Week 56
  Other Names: Beovu
  Arms: Standard regimen arm

SUMMARY:
This study is a 60-week, two-arm, randomized, open-label, active-controlled, multi-center study in patients with Polypoidal choroidal vasculopathy (PCV) who have not previously received anti-Vascular endothelial growth factor (VEGF) treatment.

DETAILED DESCRIPTION:
The purpose of this study is to measure the change in Best-corrected visual acuity (BCVA) with brolucizumab 6 mg Personalized regimen compared with Brolucizumab 6 mg Standard q12w/q8w regimen in participants with Polypoidal choroidal vasculopathy (PCV).

* The study duration will be up to 60 weeks.
* The treatment duration will be up to 56 weeks.
* The visit frequency is not fixed and may be reduced or extended depending on whether disease activity is controlled.

In the Personalized regimen arm, the first loading injection will be performed for all participants. After 4 weeks, treatment response will be judged. If there is no disease activity, injection interval will be extended to 8 weeks. The participants with presence of disease activity will continue 4-week loading injections up to 3 monthly loading dose and commence the Treat-and-extend (T&E) phase thereafter. In the T&E phase, the treatment interval can be extended by 4 weeks at a time based on Investigator's judgment of visual and/or anatomic outcomes. The maximal treatment interval is 16 weeks. At the Investigator's discretion, a participant with no disease activity or improvement of disease activity (e.g., reduction of fluid) may also be maintained on the same interval. If disease activity recurs, the interval should be shortened by 4 weeks at a time or to a minimal interval of 8 weeks.

In the Standard q12w/q8w regimen arm, all participants will receive three loading injections every 4 weeks. After loading injection, participants with no disease activity at Week 16 will receive study treatment q12w at Week 20, Week 32, and Week 44. If there is disease activity at any scheduled treatment visit, the study intervals will be adjusted to 8 weeks thereafter. Treatment intervals can be increased to 12 weeks after a treatment visit with no disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Participants ≥ 50 years of age at Screening.

   Study eye:
3. Presence of active polypoidal lesions in the macula as shown by Indocyanine green angiography (ICGA) AND presence of serosanguinous maculopathy, i.e., exudative or hemorrhagic features involving the macula on color fundus photography (CFP), Fluorescein angiography (FA) and spectral domain optical coherence tomography (SD-OCT) AND presence of Intraretinal fluid (IRF) or Subretinal fluid (SRF) that affects the central subfield as seen by SD-OCT.
4. Best-corrected visual acuity (BCVA) score must be ≤ 78 and ≥ 24 letters at 4 meters starting distance using early treatment diabetic retinopathy study (ETDRS) visual acuity charts at both Screening and Baseline.
5. Greatest liner dimension (GLD) of the total lesion area (branching vascular network [BVN] + polypoidal lesion) < 5400 μm (equivalent to 9 macular photocoagulation study [MPS] Disc Area) as delineated by Indocyanin green angiography (ICGA).

Exclusion Criteria:

Ocular conditions:

1. Concomitant conditions or ocular disorders in the study eye at Screening or Baseline which could, in the opinion of the Investigator, prevent response to study treatment or may confound interpretation of study results, compromise visual acuity or require planned medical or surgical intervention during the first 12-month study period.
2. Any active intraocular or periocular infection or active intraocular inflammation (IOI) (e.g., infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in study eye or fellow eye at Screening or Baseline.
3. Uncontrolled glaucoma in the study eye defined as intraocular pressure (IOP) > 25 mmHg on medication, or according to Investigator's judgment, at Screening or Baseline.
4. Any Polypoidal choroidal vasculopathy (PCV) masquerades like macular aneurysms, macular telangiectasia, etc. in study eye.
5. Total area of subretinal hemorrhage larger than 9 DA (Disc Area) or comprising ≥ 50% of the lesion area or presence of vitreous hemorrhage in study eye.

   Ocular treatments in the study eye:
6. Previous treatment with any anti-Vascular endothelial growth factor (VEGF) drugs or investigational drugs at any time prior to Baseline.
7. Previous use of intraocular or periocular steroids within the 6-month period prior to Baseline.
8. Macular laser photocoagulation (focal/grid) or Photodynamic therapy (PDT) at any time prior to Baseline and peripheral laser photocoagulation within 3 months prior to Baseline.

   Systemic conditions or treatments:
9. Stroke or myocardial infarction during the 6-month period prior to Baseline.
10. Systemic anti-VEGF therapy any time prior to Baseline.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Average change in Best Corrected Visual Acuity (BCVA) from Baseline at a period from Week 48 to Week 60 | from Week 48 to Week 60
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts

SECONDARY OUTCOMES:
Number of participants with last completed treatment interval of 12 weeks and/or 16-weeks with no disease activity at a period from Week 48 to Week 60 | Week 12, Week 16, and from Week 48 to Week 60
  As assessed by:
  BCVA with ETDRS charts
  Anatomical retinal evaluation of Spectral Domain Optical Coherence Tomography (SD-OCT) images
  Color fundus photography (CFP) and vascular leakage evaluation by Fluorescein angiography (FA)
  Polypoidal lesion and Branching vascular network (BVN) evaluation by Indocyanine Green Angiography (ICGA)
Distribution of last completed treatment interval with no disease activity up to Week60 | up to Week 60
  As assessed by:
  BCVA with ETDRS charts
  Anatomical retinal evaluation of Spectral Domain Optical Coherence Tomography (SD-OCT) images
  Color fundus photography (CFP) and vascular leakage evaluation by Fluorescein angiography (FA)
  Polypoidal lesion and Branching vascular network (BVN) evaluation by Indocyanine Green Angiography (ICGA)
Distribution of the maximal intervals with no disease activity up to Week 60 | up to Week 60
  As assessed by:
  BCVA with ETDRS charts
  Anatomical retinal evaluation of Spectral Domain Optical Coherence Tomography (SD-OCT) images
  Color fundus photography (CFP) and vascular leakage evaluation by Fluorescein angiography (FA)
  Polypoidal lesion and Branching vascular network (BVN) evaluation by Indocyanine Green Angiography (ICGA)
Distribution of the last interval at a period from Week 48 to Week 60 | from Week 48 to Week 60
  As assessed by:
  BCVA with ETDRS charts
  Anatomical retinal evaluation of Spectral Domain Optical Coherence Tomography (SD-OCT) images
  Color fundus photography (CFP) and vascular leakage evaluation by Fluorescein angiography (FA)
  Polypoidal lesion and Branching vascular network (BVN) evaluation by Indocyanine Green Angiography (ICGA)
Time from the last loading injection to the first visit with no disease activity | Up to Week 60
  As assessed by:
  BCVA with ETDRS charts
  Anatomical retinal evaluation of Spectral Domain Optical Coherence Tomography (SD-OCT) images
  Color fundus photography (CFP) and vascular leakage evaluation by Fluorescein angiography (FA)
  Polypoidal lesion and Branching vascular network (BVN) evaluation by Indocyanine Green Angiography (ICGA)
Occurrence of at least two successive treatment intervals with no disease activity ≥ 12-week or two successive treatment intervals with no disease activity of 16-week up to Week 60 | up to Week 60
  As assessed by:
  BCVA with ETDRS charts
  Anatomical retinal evaluation of Spectral Domain Optical Coherence Tomography (SD-OCT) images
  Color fundus photography (CFP) and vascular leakage evaluation by Fluorescein angiography (FA)
  Polypoidal lesion and Branching vascular network (BVN) evaluation by Indocyanine Green Angiography (ICGA)
Average change in BCVA from Baseline up to a period from Week 48 to Week 60 | from Week 48 to Week 60
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts
Occurrence of BCVA improvement of ≥ 10 and ≥ 15 letters from Baseline at a period from Week 48 to Week 60 | Baseline, and from Week 48 to Week 60
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts
Occurrence of BCVA ≥ 69 letters at a period from Week 48 to Week 60 | from Week 48 to Week 60
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts
Average change in BCVA from Baseline up to a period from Week 48 to Week 60 categorized into 2 groups, lower half of Baseline BCVA and upper half of Baseline BCVA | Baseline, and from Week 48 to Week 60
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts
Number of participants with complete polypoidal lesion regression at Week 12 and at a period from Week 48 to Week 60 | at Week 12, and from Week 48 to Week 60
  Polypoidal lesion and Branching vascular network (BVN) evaluation by Indocyanine Green Angiography (ICGA).
  Polypoidal regression is defined as:
  Complete polypoidal regression: complete disappearance of any hyper-cyanescent polypoidal lesion previously identified at Baseline
  Partial polypoidal regression is defined as either partial regression in number (i.e., fewer hyper-cyanescent lesions) compared with Baseline or in size (i.e., smaller hyper-cyanescent lesion) compared with Baseline
Number of participants with inactive polypoidal lesions at Week 12 and at a period from Week 48 to Week 60 | at Week 12, and from Week 48 to Week 60
  Polypoidal lesion and Branching vascular network (BVN) evaluation by Indocyanine Green Angiography (ICGA).
  Inactive polypoidal lesion is defined as the Absence of polypoidal lesions on ICGA or in case polypoidal lesions were identified or the Absence of new or persistent fluid on OCT or the Absence of leakage on angiography
Change in number and area of polypoidal lesions from Baseline at Week 12 and at a period from Week 48 to Week 60 | Baseline, Week 12, and from Week 48 to Week 60
  Polypoidal lesion and Branching vascular network (BVN) evaluation by Indocyanine Green Angiography (ICGA).
Average change from Baseline in central subfield thickness (CSFT) up to Week 60 | up to Week 60
  Change in CSFT from baseline up to week 60 will be analyzed by fitting mixed model repeated measures (MMRM) with observed data including treatment, visit, baseline central subfield thickness (CSFT) categories, age categories and treatment by visit interaction as factors.
Average change from Baseline in maximum thickness of intraretinal fluid (IRF) up to Week 60 | up to Week 60
  Change in maximum thickness of IRF from baseline up to week 60 will be analyzed by fitting mixed model repeated measures (MMRM) with observed data including treatment, visit, baseline central subfield thickness (CSFT) categories, age categories and treatment by visit interaction as factors.
Average change from Baseline in maximum thickness of subretinal fluid (SRF) up to Week 60 | up to Week 60
  Change in maximum thickness of SRF from baseline up to week 60 will be analyzed by fitting mixed model repeated measures (MMRM) with observed data including treatment, visit, baseline central subfield thickness (CSFT) categories, age categories and treatment by visit interaction as factors.
Average change from Baseline in maximum thickness of sub-retinal pigment epithelium (sub-RPE) fluid up to Week 60 | up to Week 60
  Change in maximum thickness of sub-RPE fluid from baseline up to week 60 will be analyzed by fitting mixed model repeated measures (MMRM) with observed data including treatment, visit, baseline central subfield thickness (CSFT) categories, age categories and treatment by visit interaction as factors.
Average change from Baseline in maximum thickness of pigment epithelial detachment (PED) up to Week 60 | up to Week 60
  Change in maximum PED thickness from baseline up to week 60 will be analyzed by fitting mixed model repeated measures (MMRM) with observed data including treatment, visit, baseline central subfield thickness (CSFT) categories, age categories and treatment by visit interaction as factors.
Number of participants with intraretinal fluid (IRF) and/or subretinal fluid (SRF) and/or sub-retinal pigment epithelium (sub-RPE) fluid up to Week 60 | up to Week 60
  As analyzed by fitting mixed model repeated measures (MMRM) with observed data including treatment, visit, baseline central subfield thickness (CSFT) categories, age categories and treatment by visit interaction as factors.
Incidence of ocular adverse events (AEs) up to Week 60 | Up to Week 60
  An ocular AE is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant regarding the eye.
Incidence of non-ocular adverse events (AEs) up to Week 60 | Up to Week 60
  An AE is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- South Korea (8):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Daejeon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
Access Criteria: This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/